CLINICAL TRIAL: NCT07155486
Title: A Qualitative Study on Shared Decision Making in the Choice to Use Telemonitoring in the Management of Inflammatory Bowel Disease
Brief Title: IBD-SDM Telemonitoring Interview
Status: Completed | Type: Observational
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: 2025.03.09.01
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: IBD (Inflammatory Bowel Disease); Shared Decision Making; Telemedicine; Telemonitoring
Keywords: Inflammatory Bowel Disease; Shared Decision Making
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare providers: Interviews with healthcare providers
  Interventions: Other: Interview
- Patients: Interviews with patiens
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interview

SUMMARY:
Introduction: Telemedicine has shown to play a promising role in enhancing patient care. Moreover, it is a key component of the Integraal Zorgakkoord (IZA), facilitating more efficient and accessible healthcare through telemonitoring and digital health innovations. However, it remains uncertain how Shared Decision Making (SDM) plays a role in the choice of telemedicine. Research focuses on technological capabilities or general patient-centredness, rather than how to effectively integrate SDM into decisions about using telemonitoring versus standard care. The integration of SDM into telemonitoring remains fragmented, suggesting that current SDM frameworks have not been adapted to the shift to telemedicine. If SDM is not achieved in this decision a decrease of adherence and engagement may follow.

Research question: The aim of this qualitative study is to get a better understanding of role of SDM in the choice of telemonitoring or standard care. These insights could help to offer improvements to SDM in IBD care to patients. This led to the following research questions:

1. How to optimize the decision-making process for patients with inflammatory bowel disease in the decision for telemonitoring? 1.1 How do patients and healthcare professionals perceive the current SDM within care processes for IBD?

Study design: This is a qualitative study using semi-structured interviews. Information about patient's and professionals' experiences and preferences about SDM will be collected. To guide the topics in the interview, two theories/models will be used:

1. The Three-Talk Model
2. AAMC Telehealth Competencies Data will be analysed using thematic analysis.

Study population: Consecutive adult (≥18 years) IBD patients and IBD healthcare professionals at Jeroen Bosch Hospital and Franciscus who have experienced making a choice about telemonitoring will be asked if they are willing to participate. Next, a total of 16 respondents will be include 10 patients and 6 healthcare professionals. Both patients using telemonitoring and patients who are not interested will be included. Should data saturation not have occurred, more respondents will be included.

Expected results and relevance: The objective is to investigates if and how SDM is currently integrated into the telemonitoring processes for IBD patients. The goal is to use these insights to strengthen SDM in the decision for telemonitoring for IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed IBD diagnosis

Exclusion Criteria:

* Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult (≥18 years) IBD patients and IBD healthcare professionals at JBZ and Franciscus who have experienced making a choice about telemonitoring. These hospitals are teaching institutions with a combined patient population of approximately 4000 individuals.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Explorative Data | Through study completion, an average of 2 months
  Based on topics derived from the three talk model and the AAMC Telehealth competencies. This data is evaluated with the semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Tessa EH Römkens, MD PhD, Principal Investigator — Jeroen Bosch Ziekenhuis; Rachel L West, MD PhD, Principal Investigator — Franciscus Gasthuis
Locations (2):
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Franciscus, Rotterdam

IPD SHARING:
Plan to Share IPD: No